CLINICAL TRIAL: NCT06978712
Title: Impact of Subgingival Instrumentation on Allostatic Load in Periodontitis
Brief Title: Impact of Periodontal Inflammation on Allostatic Load
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Gaytri Perio 25/35
Record Dates: First submitted 2025-05-07; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Allostatic Load; Periodontitis, Chronic
Keywords: periodontitis; inflammation; allostatic load
MeSH Terms: conditions — Chronic Periodontitis; Periodontitis; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Periodontitis (Experimental): Stage II/III Periodontitis
  Interventions: Procedure: Sub-gingival instrumentation

INTERVENTIONS:
Procedure: Sub-gingival instrumentation — All patients will undergo dental biofilm control through patient motivation, oral hygiene instructions and supragingival professional mechanical plaque removal followed by sub-gingival instrumentation.

SUMMARY:
Periodontitis is a prevalent global health issue that contributes to systemic inflammation and is closely linked to stress as a risk factor. Both conditions have been investigated for bidirectional relationship. However, the results are inconsistent, and the mechanistic links remain unclear. Allostatic load, which measures the cumulative biological effects of stress, may be relevant in elucidating this connection. Inconsistent results have been reported in previous studies exploring the association between periodontitis and individual biomarkers of allostatic load. Furthermore, none of these studies has taken into consideration staging and grading of periodontitis. Additionally, while periodontal treatment has been shown to reduce both local and systemic inflammation, its effect on allostatic load remains unexplored till date. This study aims to fill these gaps by evaluating the relationship between these parameters of periodontitis and allostatic load. Evaluation of impact of subgingival instrumentation on allostatic load may further provide insights into the broader systemic benefits of periodontal interventions.

DETAILED DESCRIPTION:
Stress is a significant risk factor for various chronic diseases, such as cardiovascular conditions, diabetes, and obesity, all of which have severe implications for public health. The relationship between stress and these chronic conditions is complex, involving both direct physiological changes and behavioural adaptations that affect health outcomes. While acute stress responses can be adaptive, chronic stress can lead to dysregulation of the body's homeostatic processes which results in allostatic load, refers to the cumulative physiological toll that the body experiences over time due to repeated or prolonged stress. Allostatic load disrupts the normal functioning of various bodily systems, including the cardiovascular, metabolic, and immune systems, which can lead to long-term health consequences such as hypertension, diabetes, and autoimmune diseases. dysregulation of the hypothalamic-pituitary-adrenal (HPA) axis and the sympathetic nervous system (SNS) during chronic stress is associated with elevated biomarkers such as cortisol, epinephrine, and dehydroepiandrosterone sulfate (DHEA-S). These biomarkers, along with other indicators like blood pressure, cholesterol, glycated haemoglobin (HbA1c), and C-reactive protein (CRP), serve as proxies for allostatic load and are critical in understanding the body's response to stress over time. Beyond its systemic effects, stress also plays a pivotal role in oral health. Chronic stress is known to increase inflammation, impair immune responses, and alter hormone levels, all of which contribute to the development and progression of oral diseases, including periodontal disease and dental caries. Stress-induced allostatic load is thought to play a role in the onset and progression of periodontal disease by disrupting the immune system and impairing the body's ability to control the microbial biofilms that contribute to the disease. Additionally, behaviours such as smoking and poor oral hygiene, which are often exacerbated by chronic stress, can further increase the risk of periodontal disease. Numerous studies have reported a bidirectional relationship between stress and periodontal disease. That is, while stress can contribute to the onset and progression of periodontal disease, the presence of periodontal disease can, in turn, exacerbate psychological stress. Despite this understanding, the exact pathogenesis of how stress affects periodontal disease remains unclear. Allostatic load provides a method for measuring the cumulative physiological effects of stress, making it a valuable tool for studying the relationship between stress and disease. This study aims to bridge this gap by examining the association between allostatic load with staging and grading of periodontitis, with a specific focus on evaluating the effects of subgingival instrumentation on allostatic load in patients with periodontitis. By addressing this critical gap in the literature, this research will contribute to a more comprehensive understanding of the interconnectedness of oral and systemic health and offer new avenues for improving patient care.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age group 30-50 years diagnosed with generalized periodontitis.
* Presence of minimum 20 teeth excluding third molars.

Exclusion Criteria:

* Periodontal treatment within last 6 months
* History of antibiotic use within the previous 3 months
* History of use of steroid, immunosuppressive and psychiatric drugs
* Pregnant and lactating women
* History of substance abuse

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 112 (Estimated)
Dates: Start 2025-06-10 (Estimated); Primary Completion 2026-06-10 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
C- Reactive protein | Baseline, 3 months
  It measures the level of inflammation in the body. Elevated CRP levels indicate infection, inflammation or disease.
HbA1c(glycated hemoglobin) | baseline, 3 months
  It measures the average level of glucose attached to hemoglobin in red blood cells over the past 2-3 months.
High Density Lipoprotein | baseline, 3 months
  It measures the amount of high density lipoprotein cholesterol level in the blood, with lower levels indicating a higher score.
Bleeding on Probing | Baseline, 3 months
  It will be recorded as bleeding occurring within 15 seconds of probing.

CONTACTS AND LOCATIONS:
Locations (1):
- PGIDS, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No